CLINICAL TRIAL: NCT06786312
Title: A Single-arm, Multicenter, Prospective Phase II Clinical Study of Apatinib in Combination With Adebrelimab and EC Regimen in the First-line Treatment of Extensive Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG 010
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: Adebrelimab; Apatinib; EC; Small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Apatinib; Drug: Adebrelimab; Drug: Etoposide Injection; Drug: Carboplatin Injection

INTERVENTIONS:
Drug: Apatinib — 250mg, P.O, qd, 21 days per cycle;
Drug: Adebrelimab — 20mg/kg or 1200mg ivgtt, d1, 21 days per cycle;
Drug: Etoposide Injection — 100mg/m^2 ivgtt for the first, second and third consecutive days, 21 days per cycle.
Drug: Carboplatin Injection — Day 1 administration, AUC=5, intravenous infusion; One treatment cycle every 21 days.

SUMMARY:
To evaluate the efficacy and safety of apatinib combined with adebrelizumab and EC in the first-line treatment of extensive small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with extensive stage small cell lung cancer confirmed by histopathology or cytology (excluding complex small cell lung cancer);
* 2. Age at the time of signing the informed consent: 18-75 years old (including 18 and 75 years old), male or female;
* 3. The physical status of the Eastern Oncology Consortium (ECOG) was 0 or 1 (see Annex 1 for the ECOGPS scoring criteria);
* 4. Have not received systematic treatment for extensive small cell lung cancer;
* 5. Have at least one measurable lesion that meets the RECIST v1.1 standard (see Annex 3);
* 6. Expected survival >=3 months;
* 7. If the major organs function normally, the following criteria are met:

  1. Blood routine test: hemoglobin (Hb) >=90g/L; Absolute neutrophil count (ANC) >=1.5×10^9/L; Platelet (PLT) >=100×10^9/L; White blood cell count (WBC) >= 3.0×10^9/L;
  2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=2.5×ULN (tumor liver metastasis, <=5×ULN); Serum total bilirubin (TBIL) <=1.5×ULN (Gilbert syndrome subjects, <=3×ULN; In patients with liver metastasis, total bilirubin <=3× ULN); Serum creatinine (Cr) <=1.5×ULN or creatinine clearance >=50ml/min;
  3. Coagulation function: activated partial thromboplastin time (APTT), International standardized ratio (INR), prothrombin time (PT) <=1.5×ULN;
  4. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF)>=50%;
* 8. BMS must be asymptomatic or treated and stable after discontinuation of steroids and anticonvulsants for at least 1 month prior to study therapy;
* 9. Women of reproductive age should agree that they must use contraceptives (such as intrauterine devices [IUD], birth control pills or condoms) during the study period and for 6 months after the study ends; Have a negative serum pregnancy test within 28 days prior to study enrollment and must be a non-lactating subject; Men should be subjects who agree to use contraception during the study period and for 6 months after the end of the study period.
* 10. Subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* 1. Known allergy to any of the drugs in the study;
* 2. Previous or co-existing malignancies other than cured basal cell carcinoma of the skin, cervical carcinoma in situ, ductal carcinoma in situ of the breast (DCIS), papillary carcinoma of the thyroid gland, and other malignancies that have been adequately treated and cured for ≥5 years prior to the first dose with evidence of no recurrence or metastasis;
* 3. Presence of symptomatic or active central nervous system (CNS) metastases or cancerous meningitis (patients with asymptomatic or stable brain metastases after treatment are allowed to be included);
* 4. Active or previously suffering from autoimmune disease or immune deficiency;
* 5. In the first study, patients with clinically significant bleeding symptoms or bleeding tendency, such as hemoptysis, hematemesis, hematochezia, gastrointestinal bleeding, hemorrhagic gastric ulcer, etc., occurred within 3 months before medication;
* 6. Imaging (CT or MRI) shows that the tumor has invaded the large blood vessels or the boundary with the large blood vessels is unclear; Or if the investigator determines that the subject's tumor has a high risk of invading vital blood vessels during treatment and causing fatal bleeding;
* 7. Have high blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure >= 150mmHg or diastolic blood pressure >= 100 mmHg);
* 8. Cardiovascular and cerebrovascular diseases of significant clinical significance:

  1. Cerebrovascular accident (excluding lacunar infarction, minor cerebral ischemia, or transient ischemic attack), myocardial infarction, unstable angina pectoris, and poorly controlled arrhythmias (including QTc interval >= 450ms for men and 470 ms for women) occurred within 6 months before the first administration of the study drug (QTc interval >= 450ms for women) Fridericia formula);
  2. New York Heart Association (NYHA) heart function Grade > II or left ventricular ejection fraction (LVEF) < 50%;
* 9. Active or uncontrolled severe infection;

  1. Known human immunodeficiency virus (HIV) infection;
  2. Known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., HBV DNA positive (>1×104 copies /mL or >2000 IU/ml) must be excluded for a known HBV carrier;
  3. Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis;
* 10. Patients with uncontrolled pleural effusion, pericardial effusion or peritoneal effusion in the third space, as judged by researchers, requiring puncture and drainage; Or received ascites, pleural effusion drainage within 14 days before the first medication;
* 11. Patients with interstitial pneumonia or interstitial lung disease, or a history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other pulmonary fibrosis, chronic pneumonia, pneumonia due to drug or radiation therapy, a history of congenital pneumonia, or any evidence of active pneumonia on chest CT scan that may interfere with the judgment of immune-related pulmonary toxicity; Patients with severe impairment of lung function confirmed by current pulmonary function examination;
* 12. Subjects who required systemic corticosteroids (> 10 mg/ day effective dose of prednisone) or other immunosuppressive agents within 14 days prior to initial dosing or during the study period. However, in the absence of active autoimmune disease, subjects were allowed to receive topical or inhaled steroids and adrenal hormone replacement therapy at a dose <=10 mg/ day of prednisone effectiveness;
* 13. The subject has any current disease or condition that affects drug absorption, or the subject is unable to take apatinib orally;
* 14. Urine routine indicated urinary protein >=2+, and 24-hour urinary protein quantity >1.0g;
* 15. The investigator considers that the subject is not suitable to participate in the clinical study due to any clinical or laboratory abnormalities or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2027-07-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 0ne year
  Defined as the time from the start of enrollment to the date when objective tumor progression was first recorded or to death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective remission rate | one year
  Proportion of subjects with CR and PR (RECIST v1.1 standard)
Disease control rate | one year
  Proportion of subjects with CR and PR and SD (RECIST v1.1 standard)
Overall survival | 2 years
  Defined as the time between enrollment and the subject's death from various causes;
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fuzhou

IPD SHARING:
Plan to Share IPD: Undecided